CLINICAL TRIAL: NCT03376841
Title: An Open-Label Study to Evaluate the Effect of Severe Hepatic Impairment on the Pharmacokinetics of Cenicriviroc and Its Metabolites Following Single Dose Administration
Brief Title: Impact of Severe Hepatic Impairment on Pharmacokinetics of Cenicriviroc and Its Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3152-102-002
Record Dates: First submitted 2017-08-02; First posted 2017-12-19 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Hepatic Impairment
Keywords: Liver insufficiency; Hepatic Impairment; Cenicriviroc; Pharmacokinetics
MeSH Terms: conditions — Hepatic Insufficiency | interventions — cenicriviroc

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe hepatic impairment (Experimental): Cenicriviroc tablet; single-dose oral administration
  Interventions: Drug: Cenicriviroc
- Normal Hepatic function (Experimental): Cenicriviroc tablet; single-dose oral administration
  Interventions: Drug: Cenicriviroc

INTERVENTIONS:
Drug: Cenicriviroc — 1 tablet; single-dose oral administration
  Other Names: CVC

SUMMARY:
The objective of this study is to assess the pharmacokinetics (PK), safety, and tolerability profiles of cenicriviroc (CVC) and its metabolites (M-I and M-II) in participants with severely impaired hepatic function compared with matched healthy participants following single-dose administration

ELIGIBILITY:
Inclusion Criteria for all participants:

* Sign the ICF and have the mental capability to understand it
* If female, have a negative result from a serum pregnancy test at screening and a negative result from a serum or urine pregnancy test on Day -1
* If male, agree to use an effective method of contraception (ie, condom plus diaphragm with spermicide or condom plus spermicide) and not have their partners become pregnant for at least 30 days after dosing study treatment, or have been sterilized for at least 1 year
* If female of childbearing potential, agree to use an effective method of contraception (ie, condom plus diaphragm with spermicide, condom plus spermicide, or nonhormonal intrauterine device) and not become pregnant for at least 30 days after dosing study treatment. Females who are at least 2 years postmenopausal (with supporting documentation from an obstetrician/gynecologist) or who have had tubal ligation or hysterectomy (with supporting documentation from the physician who performed the surgery) will not be considered to be of childbearing potential
* Be nonsmoking (never smoked or have not smoked in the previous 2 years) or a light smoker (fewer than 10 cigarettes per day within 1 week prior to study treatment administration)
* Have a body mass index (BMI) ≥ 18 kg/m2 and ≤ 42 kg/m2

Inclusion Criteria for Participants with Severely Impaired Hepatic Function:

* Have chronic liver disease and/or cirrhosis documented by the presence of at least 1 of the following:

  1. Liver biopsy with histologic findings consistent with cirrhosis
  2. Computerized tomographic or ultrasonographic evidence of liver disease with or without portal hypertension
  3. Physical examination and clinical and laboratory evidence of chronic liver disease
  4. Colloid shift on a liver-spleen scan

     Exclusion Criteria for all participants:
* Known hypersensitivity to cenicriviroc and other chemokine receptor 2 and/or 5 (CCR2 and/or CCR5) antagonists such as maraviroc (CCR5 antagonist)
* History of substance abuse within the previous 2 years
* Dosing in any other clinical investigation using an experimental drug requiring repeated blood or plasma draws within 30 days of study treatment administration
* Participation in a blood or plasma donation program within 60 or 30 days, respectively, of study treatment administration
* Consumption of caffeine within 48 hours prior to dosing; consumption of grapefruit containing products, vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), foods containing poppy seeds, and charbroiled meats within 14 days prior to dosing; or consumption of alcohol within 72 hours prior to dosing before study treatment administration
* Employee, or immediate relative of an employee, of the sponsor, any of its affiliates or partners, or the study center
* Previously taken cenicriviroc or previously participated in an investigational study of cenicriviroc
* Pregnant or breastfeeding (female participants)

Exclusion Criteria for Participants with Severely Impaired Hepatic Function:

* Have an acute exacerbation of liver disease as indicated by worsening clinical signs and/or laboratory tests within the 4 weeks before study treatment administration
* Have ascites that will require paracentesis within 1 week of dosing or during the study period
* Have gastrointestinal hemorrhage due to esophageal varices, peptic ulcers or Mallory Weiss Syndrome within 6 months before Day 1, unless banded and stable
* Have a Child-Pugh score of < 10
* Any clinical condition other than hepatic impairment or previous surgery that might affect the absorption, distribution, biotransformation, or excretion of cenicriviroc and its metabolites

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) from time 0 to time t (AUC0-t) | 6 days (144 hours)
AUC from time 0 to infinity (AUC0-∞) | 6 days (144 hours)
Maximum plasma drug concentration (Cmax) | 6 days (144 hours)

SECONDARY OUTCOMES:
Time of maximum plasma drug concentration (Tmax) | 6 days (144 hours)
Terminal elimination rate constant | 6 days (144 hours)
Terminal elimination half-life (T½) | 6 days (144 hours)
Total body clearance of drug from plasma (CL/F for CVC only) | 6 days (144 hours)
Volume of distribution during the terminal phase (Vz/F for CVC only) | 6 days (144 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Surya Ayalasomayajula, Study Director — Allergan
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com